CLINICAL TRIAL: NCT01600885
Title: The Effects of Ketamine and Guanfacine on Working Memory in Healthy Subjects
Acronym: GuaKet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0807004092
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: NMDA Receptor Function
Keywords: Guanfacine; Ketamine; Functional Magnetic Resonance Imaging; Prefrontal Cortex Activity; Receptors, N-Methyl-D-Aspartate; Receptors, Adrenergic, alpha-2; Memory, Short-Term; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guanfacine then Placebo (Active Comparator): During the first study session, the participant will receive guanfacine before undergoing a ketamine-infusion fMRI. During the second study session, at least two weeks later, the participant will receive a placebo before undergoing a ketamine-infusion fMRI.
  Interventions: Drug: Guanfacine; Drug: Placebo
- Placebo then Guanfacine (Active Comparator): During the first study session, the participant will receive a placebo before undergoing a ketamine-infusion fMRI. During the second study session, at least two weeks later, the participant will receive guanfacine before undergoing a ketamine-infusion fMRI.
  Interventions: Drug: Guanfacine; Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — Subjects will be given 3mg of guanfacine before the fMRI scan. Then when in the scanner, a bolus of ketamine (0.23mg/kg over 1 min) will be given during the visual fixation scan. Immediately after completion of the 1 min bolus, the participant will receive a steady state ketamine infusion of 0.58 mg/kg/hour and brain activation will be measured during a spatial working memory task. The entire scan will last approximately two and a half hours and the ketamine infusion will be up to one hour and 15 minutes.
Drug: Placebo — Subjects will be given a placebo before the fMRI scan. Then when in the scanner, a bolus of ketamine (0.23mg/kg over 1 min) will be given during the visual fixation scan. Immediately after completion of the 1 min bolus, the participant will receive a steady state ketamine infusion of 0.58 mg/kg/hour and brain activation will be measured during a spatial working memory task. The entire scan will last approximately two and a half hours and the ketamine infusion will be up to one hour and 15 minutes.

SUMMARY:
The purpose of the study is

1. To establish the feasibility of fMRI studies of the interaction of guanfacine and ketamine.
2. To explore the possibility that guanfacine can ameliorate the negative effects of ketamine on task-related prefrontal activation.
3. To assess the strength of any interaction between guanfacine and ketamine.

DETAILED DESCRIPTION:
Potential subjects will be interviewed over the phone and, if appropriate, will be scheduled for a screening session. Participants who meet study criteria will participate in two study sessions separated by at least two weeks. The sessions will be identical except on one day they will receive guanfacine and on the other, they will receive a placebo.

This study was initially completed in 2014. Upon analysis of the collected data, it was decided to add additional subjects and gather additional data to verify results seen in the collected data. The study was reopened and new data was added beginning in September 2016. Information about the study beginning in 2016 is available in a separate record.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 45, inclusive
* Right-handed
* Have at least a 12th grade education level or equivalent
* Able to read and write English as a primary language
* Willing to refrain from caffeine and alcohol use for one week prior to each MRI session.

Exclusion Criteria:

* Abnormality on physical examination
* A 12 lead ECG at screening has clinically significant abnormalities as determined by the physician reading the ECG
* A positive pre-study urine drug screen or, at the study physicians' discretion on any drug screens given before the scans
* Abnormality on clinical chemistry or hematology examination at the pre-study medical screening.
* History of positive HIV or Hepatitis B.
* Has received either prescribed or over-the-counter (OTC) centrally active medicine or herbal supplements within the week prior to the MRI scan.
* History of any substance abuse disorder meeting DSM-IV criteria with the exception of nicotine
* Any history of DSM-IV Axis I psychiatric disorders,
* Any history of major medical or neurological disorders
* Any history indicating learning disability, mental retardation, or attention deficit disorder.
* First-degree relative with Axis I DSM-IV disorder including substance abuse or dependence.
* Any clinically significant abnormalities on screening electrocardiogram
* Any history of head injury
* Any evidence of psychosis-like symptoms, as indicated by elevated scores on the Perceptual Aberration-Magical Ideation (Chapman, Chapman et al. 1978; Eckblad, Chapman et al. 1983) and the revised Social Anhedonia scales(Eckblad, Chapman et al. unpublished)
* A positive urine toxicology screen for illicit substance use or positive alcohol breathalyzer test conducted at screening interview and prior to each MRI session
* Known sensitivity to ketamine.
* Body circumference of 52 inches or greater.
* History of claustrophobia
* Any clinically significant impairment of color vision or visual acuity after correction available in the scanner.
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI screening questionnaire
* Pregnancy or breast-feeding would exclude potential participants and all female subjects will receive a urine pregnancy test at screening and before each MRI scan.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Blood pressure must be higher than 90/70. Pulse must be greater than 40 unless the participant is cleared by a study physician

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Krystal, M.D., Principal Investigator — Yale University; Naomi R Driesen, Ph.D., Study Director — Yale University
Locations (3):
- United States (3):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale Magnetic Resonance Research Center, New Haven, Connecticut
  - Veterans Affairs Hospital, West Haven, Connecticut

REFERENCES:
- [Background] Arnsten AF, Cai JX. Postsynaptic alpha-2 receptor stimulation improves memory in aged monkeys: indirect effects of yohimbine versus direct effects of clonidine. Neurobiol Aging. 1993 Nov-Dec;14(6):597-603. doi: 10.1016/0197-4580(93)90044-c. PMID 7905189
- [Background] Bjarnadottir M, Misner DL, Haverfield-Gross S, Bruun S, Helgason VG, Stefansson H, Sigmundsson A, Firth DR, Nielsen B, Stefansdottir R, Novak TJ, Stefansson K, Gurney ME, Andresson T. Neuregulin1 (NRG1) signaling through Fyn modulates NMDA receptor phosphorylation: differential synaptic function in NRG1+/- knock-outs compared with wild-type mice. J Neurosci. 2007 Apr 25;27(17):4519-29. doi: 10.1523/JNEUROSCI.4314-06.2007. PMID 17460065
- [Background] Brandt, J. The Hopkins Verbal Learning Test: development of a new memory test with six equivalent forms The Clinical Neuropsychologist 125-142, 1991
- [Background] Buccafusco JJ. Neuropharmacologic and behavioral actions of clonidine: interactions with central neurotransmitters. Int Rev Neurobiol. 1992;33:55-107. doi: 10.1016/s0074-7742(08)60691-1. No abstract available. PMID 1350577
- [Background] Chapman LJ, Chapman JP, Raulin ML. Body-image aberration in Schizophrenia. J Abnorm Psychol. 1978 Aug;87(4):399-407. doi: 10.1037//0021-843x.87.4.399. No abstract available. PMID 681612
- [Background] Cho HS, D'Souza DC, Gueorguieva R, Perry EB, Madonick S, Karper LP, Abi-Dargham A, Belger A, Abi-Saab W, Lipschitz D, Bennet A, Seibyl JP, Krystal JH. Absence of behavioral sensitization in healthy human subjects following repeated exposure to ketamine. Psychopharmacology (Berl). 2005 Apr;179(1):136-43. doi: 10.1007/s00213-004-2066-5. Epub 2005 Jan 29. PMID 15682309
- [Background] da Silva TL, Pianca TG, Roman T, Hutz MH, Faraone SV, Schmitz M, Rohde LA. Adrenergic alpha2A receptor gene and response to methylphenidate in attention-deficit/hyperactivity disorder-predominantly inattentive type. J Neural Transm (Vienna). 2008;115(2):341-5. doi: 10.1007/s00702-007-0835-0. Epub 2008 Jan 16. PMID 18200436
- [Background] Driesen NR, Leung HC, Calhoun VD, Constable RT, Gueorguieva R, Hoffman R, Skudlarski P, Goldman-Rakic PS, Krystal JH. Impairment of working memory maintenance and response in schizophrenia: functional magnetic resonance imaging evidence. Biol Psychiatry. 2008 Dec 15;64(12):1026-34. doi: 10.1016/j.biopsych.2008.07.029. Epub 2008 Sep 27. PMID 18823880
- [Background] Eckblad M, Chapman LJ. Magical ideation as an indicator of schizotypy. J Consult Clin Psychol. 1983 Apr;51(2):215-25. doi: 10.1037//0022-006x.51.2.215. No abstract available. PMID 6841765
- [Background] Friedman JI, Adler DN, Temporini HD, Kemether E, Harvey PD, White L, Parrella M, Davis KL. Guanfacine treatment of cognitive impairment in schizophrenia. Neuropsychopharmacology. 2001 Sep;25(3):402-9. doi: 10.1016/S0893-133X(01)00249-4. PMID 11522468
- [Background] Glantz LA, Lewis DA. Dendritic spine density in schizophrenia and depression. Arch Gen Psychiatry. 2001 Feb;58(2):203. doi: 10.1001/archpsyc.58.2.203. No abstract available. PMID 11177126
- [Background] Glantz LA, Lewis DA. Decreased dendritic spine density on prefrontal cortical pyramidal neurons in schizophrenia. Arch Gen Psychiatry. 2000 Jan;57(1):65-73. doi: 10.1001/archpsyc.57.1.65. PMID 10632234
- [Background] Hahn CG, Wang HY, Cho DS, Talbot K, Gur RE, Berrettini WH, Bakshi K, Kamins J, Borgmann-Winter KE, Siegel SJ, Gallop RJ, Arnold SE. Altered neuregulin 1-erbB4 signaling contributes to NMDA receptor hypofunction in schizophrenia. Nat Med. 2006 Jul;12(7):824-8. doi: 10.1038/nm1418. Epub 2006 Jun 11. PMID 16767099
- [Background] Hunt RD, Arnsten AF, Asbell MD. An open trial of guanfacine in the treatment of attention-deficit hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 1995 Jan;34(1):50-4. doi: 10.1097/00004583-199501000-00013. PMID 7860456
- [Background] Jakala P, Riekkinen M, Sirvio J, Koivisto E, Kejonen K, Vanhanen M, Riekkinen P Jr. Guanfacine, but not clonidine, improves planning and working memory performance in humans. Neuropsychopharmacology. 1999 May;20(5):460-70. doi: 10.1016/S0893-133X(98)00127-4. PMID 10192826
- [Background] Kaye, S., L. Opler, et al. (1986) Positive and Negative Syndrome Scale. Toronto, Ontario. Multi-Health Systems, Inc.
- [Background] Kirkpatrick B, Xu L, Cascella N, Ozeki Y, Sawa A, Roberts RC. DISC1 immunoreactivity at the light and ultrastructural level in the human neocortex. J Comp Neurol. 2006 Jul 20;497(3):436-50. doi: 10.1002/cne.21007. PMID 16736468
- [Background] Krystal JH, Perry EB Jr, Gueorguieva R, Belger A, Madonick SH, Abi-Dargham A, Cooper TB, Macdougall L, Abi-Saab W, D'Souza DC. Comparative and interactive human psychopharmacologic effects of ketamine and amphetamine: implications for glutamatergic and dopaminergic model psychoses and cognitive function. Arch Gen Psychiatry. 2005 Sep;62(9):985-94. doi: 10.1001/archpsyc.62.9.985. PMID 16143730
- [Background] Leung HC, Gore JC, Goldman-Rakic PS. Sustained mnemonic response in the human middle frontal gyrus during on-line storage of spatial memoranda. J Cogn Neurosci. 2002 May 15;14(4):659-71. doi: 10.1162/08989290260045882. PMID 12126506
- [Background] Ma CL, Arnsten AF, Li BM. Locomotor hyperactivity induced by blockade of prefrontal cortical alpha2-adrenoceptors in monkeys. Biol Psychiatry. 2005 Jan 15;57(2):192-5. doi: 10.1016/j.biopsych.2004.11.004. PMID 15652880
- [Background] McClure MM, Barch DM, Romero MJ, Minzenberg MJ, Triebwasser J, Harvey PD, Siever LJ. The effects of guanfacine on context processing abnormalities in schizotypal personality disorder. Biol Psychiatry. 2007 May 15;61(10):1157-60. doi: 10.1016/j.biopsych.2006.06.034. Epub 2006 Sep 1. PMID 16950221
- [Background] Newcomer, J., N. Farber, et al. (1999).
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Polanczyk G, Zeni C, Genro JP, Guimaraes AP, Roman T, Hutz MH, Rohde LA. Association of the adrenergic alpha2A receptor gene with methylphenidate improvement of inattentive symptoms in children and adolescents with attention-deficit/hyperactivity disorder. Arch Gen Psychiatry. 2007 Feb;64(2):218-24. doi: 10.1001/archpsyc.64.2.218. PMID 17283289
- [Background] Small KM, Brown KM, Seman CA, Theiss CT, Liggett SB. Complex haplotypes derived from noncoding polymorphisms of the intronless alpha2A-adrenergic gene diversify receptor expression. Proc Natl Acad Sci U S A. 2006 Apr 4;103(14):5472-7. doi: 10.1073/pnas.0601345103. Epub 2006 Mar 27. PMID 16567612
- [Background] Swartz BE, Kovalik E, Thomas K, Torgersen D, Mandelkern MA. The effects of an alpha-2 adrenergic agonist, guanfacine, on rCBF in human cortex in normal controls and subjects with focal epilepsy. Neuropsychopharmacology. 2000 Sep;23(3):263-75. doi: 10.1016/S0893-133X(00)00101-9. PMID 10942850
- [Background] Szabo B. Imidazoline antihypertensive drugs: a critical review on their mechanism of action. Pharmacol Ther. 2002 Jan;93(1):1-35. doi: 10.1016/s0163-7258(01)00170-x. PMID 11916539
- [Background] Wang M, Ramos BP, Paspalas CD, Shu Y, Simen A, Duque A, Vijayraghavan S, Brennan A, Dudley A, Nou E, Mazer JA, McCormick DA, Arnsten AF. Alpha2A-adrenoceptors strengthen working memory networks by inhibiting cAMP-HCN channel signaling in prefrontal cortex. Cell. 2007 Apr 20;129(2):397-410. doi: 10.1016/j.cell.2007.03.015. PMID 17448997
- [Background] Wang Q, Jaaro-Peled H, Sawa A, Brandon NJ. How has DISC1 enabled drug discovery? Mol Cell Neurosci. 2008 Feb;37(2):187-95. doi: 10.1016/j.mcn.2007.10.006. Epub 2007 Oct 23. PMID 18055216

RESULTS

PARTICIPANT FLOW:
Groups:
- Guanfacine Then Placebo: During the first study session, the participant will receive guanfacine before undergoing a ketamine-infusion fMRI. During the second study session, at least two weeks later, the participant will receive a placebo before undergoing a ketamine-infusion fMRI.
  Guanfacine then Placebo: During the first study session, the patient will be given 3mg of guanfacine before the fMRI scan. Then when in the scanner, a bolus of ketamine (0.23mg/kg over 1 min) will be given during the visual fixation scan. Immediately after completion of the 1 min bolus, the participant will receive a steady state ketamine infusion of 0.58 mg/kg/hour and brain activation will be measured during a spatial working memory task. The entire scan will last approximately two and a half hours and the ketamine infusion will be up to one hour and 15 minutes.
  The second study session will be identical except that the patient will be given a placebo instead of the guanfacine.
- Placebo Then Guanfacine: During the first study session, the participant will receive a placebo before undergoing a ketamine-infusion fMRI. During the second study session, at least two weeks later, the participant will receive guanfacine before undergoing a ketamine-infusion fMRI.
  Placebo then Guanfacine: During the first study session, the patient will be given a placebo before the fMRI scan. Then when in the scanner, a bolus of ketamine (0.23mg/kg over 1 min) will be given during the visual fixation scan. Immediately after completion of the 1 min bolus, the participant will receive a steady state ketamine infusion of 0.58 mg/kg/hour and brain activation will be measured during a spatial working memory task. The entire scan will last approximately two and a half hours and the ketamine infusion will be up to one hour and 15 minutes.
  The second study session will be identical except that the patient will be given 3mg of guanfacine instead of the placebo.
Period: First Period
Arm/Group | Guanfacine Then Placebo | Placebo Then Guanfacine
Started | 10 | 9
Completed | 8 | 8
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — moved out of area | 1 | 0
Period: Wash Out Period
Arm/Group | Guanfacine Then Placebo | Placebo Then Guanfacine
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Period
Arm/Group | Guanfacine Then Placebo | Placebo Then Guanfacine
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population is the number of participants who started the study
Groups:
- Overall Study: This 'arm' consists of all study participants who started the first Study Period. This Study Period consisted of an initial screening visit in which it was determined whether participants met the inclusion/exclusion criteria for further participation in this study.
Arm/Group | Overall Study
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Amelioration of Ketamine-related Task Activation as Measured by Functional Magnetic Resonance Imaging in Inferior Parietal Lobule
Description: Scans will be analyzed for task-related prefrontal activation
  Difference Score: Percent Signal Change in Regions of Interest (ketamine - saline)
Time Frame: Within 4 hours of dose administration, after up to 1.25 hours of ketamine infusion
Population: ALL SUBJECTS WHO COMPLETED THE STUDY WERE INCLUDED IN ANALYSIS
Measure: Mean (Standard Error); unit: percent change in saline signal
Groups:
- Guanfacine: Subjects were given 3mg of guanfacine before the fMRI scan. Then when in the scanner, a bolus of ketamine (0.23mg/kg over 1 min) was given during the visual fixation scan. Immediately after completion of the 1 min bolus, the subjects received a steady state ketamine infusion of 0.58 mg/kg/hour and brain activation was measured during a spatial working memory task. The entire scan lasted approximately two and a half hours and the ketamine infusion lasted up to one hour and 15 minutes.
- Placebo: Subjects were given a placebo before the fMRI scan. Then when in the scanner, a bolus of ketamine (0.23mg/kg over 1 min) was given during the visual fixation scan. Immediately after completion of the 1 min bolus, the participant received a steady state ketamine infusion of 0.58 mg/kg/hour and brain activation was measured during a spatial working memory task. The entire scan lasted approximately two and a half hours and the ketamine infusion lasted up to one hour and 15 minutes.
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 16 | 16
percent change in saline signal | -0.17 (0.046) | -0.094 (0.054)

2. Primary Outcome: Percent Change in Amelioration of Ketamine-related Task Activation as Measured by Functional Magnetic Resonance Imaging in Middle Frontal Gyrus
Description: Difference Score: Percent Signal Change in Regions of Interest (ketamine - saline)
Time Frame: Within 4 hours of dose administration, after up to 1.25 hours of ketamine infusion
Population: ALL SUBJECTS WHO COMPLETED THE STUDY WERE INCLUDED IN ANALYSIS
Measure: Mean (Standard Error); unit: percent change in saline signal
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 16 | 16
percent change in saline signal | -0.1 (0.052) | 0.052 (0.0652)

3. Primary Outcome: Percent Change in Amelioration of Ketamine-related Task Activation as Measured by Functional Magnetic Resonance Imaging in Superior Frontal Gyrus
Description: Difference Score: Percent Signal Change in Regions of Interest (ketamine - saline)
Time Frame: Within 4 hours of dose administration, after up to 1.25 hours of ketamine infusion
Population: ALL SUBJECTS WHO COMPLETED THE STUDY WERE INCLUDED IN ANALYSIS
Measure: Mean (Standard Error); unit: percent change in saline signal
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 16 | 16
percent change in saline signal | -0.134 (0.0413) | -0.086 (0.0365)

ADVERSE EVENTS:
Time Frame: Throughout the length of the study (Aproximately 3 years)
Groups:
- Placebo: Subjects were given 3mg of guanfacine before the fMRI scan. Then when in the scanner, a bolus of ketamine (0.23mg/kg over 1 min) was given during the visual fixation scan. Immediately after completion of the 1 min bolus, the subjects received a steady state ketamine infusion of 0.58 mg/kg/hour and brain activation was measured during a spatial working memory task. The entire scan lasted approximately two and a half hours and the ketamine infusion lasted up to one hour and 15 minutes.
Arm/Group | Guanfacine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No